CLINICAL TRIAL: NCT06580899
Title: Effectiveness of Continuous Local Infiltration Analgesia Intra-Articular Catheters for Pain Relief in Total Knee Replacement
Brief Title: Intra-Articular Catheter Total Knee Arthroplasty
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CONC005
Record Dates: First submitted 2024-08-08; First posted 2024-08-30 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Continuous Local Infiltration Analgesia; Intra-articular Catheter; Total Knee Arthroplasty
Keywords: continuous local infiltration analgesia; intra-articular catheter
MeSH Terms: interventions — Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- No post-operative intra-articular catheter (Other): Subjects that receive ONLY the existing standard of care (SOC) multimodal pain management protocol and DO NOT receive post-operative intra-articular catheter.
  Interventions: Other: Routine Standard of Care Treatment
- BRAND 1 intra-articular catheter (Active Comparator): Subjects that receive the BRAND 1 intra-articular catheter pump with existing SOC multimodal pain management protocol in the immediate post-op period.
  Interventions: Device: Intra-articular catheter
- BRAND 2 intra-articular catheter (Active Comparator): Subjects that receive the newer BRAND 2 intra-articular catheter pump with existing SOC multimodal pain management protocol in the immediate post-op period.
  Interventions: Device: Intra-articular catheter

INTERVENTIONS:
Device: Intra-articular catheter — Intra-articular catheter pump with existing standard-of-care multimodal pain management protocol in the immediate post-op period
  Arms: BRAND 1 intra-articular catheter; BRAND 2 intra-articular catheter
Other: Routine Standard of Care Treatment — No changes to what would occur outside of the study.
  Arms: No post-operative intra-articular catheter

SUMMARY:
This is a prospective, randomized clinical trial evaluating three groups. The groups are:

Group 1 (Control): Subjects that receive only the existing standard-of-care multimodal pain management protocol and do not receive post-operative intra-articular catheter.

Group 2 (Investigational Treatment/Intervention): Subjects that receive the brand 1 intra-articular catheter pump with existing standard-of-care multimodal pain management protocol in the immediate post-operative period.

Group 3 (Investigational Treatment/Intervention): Subjects that receive the newer brand 2 intra-articular catheter pump with existing standard-of-care multimodal pain management protocol in the immediate post-operative period.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effects of one of two continuous local infiltration analgesia (intra-articular catheter device) on patient postoperative pain scores following primary unilateral total knee arthroplasty in comparison to no addition of an intra-articular (IART) catheter post total knee arthroplasty (TKA). The investigators hypothesize that if patients undergoing primary unilateral TKA surgery receive an intra-articular catheter device that continuously delivers local infiltration analgesia in the postoperative period, then their postoperative pain scores on the visual analog scale will decrease. Secondary objectives will include determining the role of intraoperative tourniquet use on thigh versus knee postoperative pain and quantifying the amount of additional postoperative patient communication related to the intra-articular catheter device.

Previous literature demonstrates conflicting results on the effects of continuous local infiltration analgesia on postoperative pain management following TKA. The proposed study incorporates a well-designed and substantially powered study to directly compare patient postoperative pain scores with and without the use of an intra-articular catheter device, which will provide additional evidence and clarity to the literature.

If the intra-articular catheter is determined to provide meaningful reductions in postoperative pain, this directly benefits patients undergoing TKA surgery. Decreases in postoperative pain allow for increased patient comfort and earlier functional knee rehabilitation following surgery, both of which promote a faster recovery. A favorable intra-articular catheter study, in addition to the previous literature on continuous local infiltration analgesia, has the potential to change the previous standard of care following TKA surgery to add intra-articular catheter or similar devices as an evidence-based treatment in multimodal pain protocols. If the intra-articular catheter is determined not to provide clinically significant reductions in postoperative pain, then these devices have no substantial benefit to the patient and orthopedic surgeons can stop prescribing them. TKA surgery would become more cost-effective as the additional cost associated with the intra-articular catheter device will no longer be charged. The intraarticular intra-articular catheter patient pump has a rare, but small risk of infection due to the portal from the external environment to the knee joint. This additional catheter infection risk will be eliminated if future use of the intra-articular catheter device subsides.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective outpatient unilateral TKA at Mallard Creek Surgery Center
2. Subjects ≥ 18 years or age
3. Subjects willing and able to provide written informed consent to participate in this study
4. Subjects who are indicated to use an intra-articular catheter pump system

Exclusion Criteria:

1. Subjects < 18 years of age
2. Subjects with history of chronic pain, neuropathic pain, or currently enrolled in pain management agreement
3. Subjects undergoing bilateral TKA
4. Subjects taking opiate pain medication preoperatively within 6 weeks of surgery date.
5. Subjects allergic to any components or treatment medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 2 days postoperative, 2 weeks postoperative
  Numeric Pain Rating Scale (0-10 scale where 10 is worse)

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS Jr.) | 6 weeks postoperative
  KOOS Jr. The interval score ranges from 0 to 100 where 0 represents total knee disability and 100 represents perfect knee health

OTHER OUTCOMES:
Anesthesia Type | at time of surgery
  type of anesthesia used during procedure
tourniquet times | at time of surgery
  how long was a tourniquet used during procedure
range of motion | preoperative, 2 weeks postoperative, 6 weeks postoperative
  knee range of motion

CONTACTS AND LOCATIONS:
Locations (1):
- OrthoCarolina Research Institute, Inc., Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No IPD sharing

REFERENCES:
- [Background] Gunaratne R, Pratt DN, Banda J, Fick DP, Khan RJK, Robertson BW. Patient Dissatisfaction Following Total Knee Arthroplasty: A Systematic Review of the Literature. J Arthroplasty. 2017 Dec;32(12):3854-3860. doi: 10.1016/j.arth.2017.07.021. Epub 2017 Jul 21. PMID 28844632
- [Background] Li JW, Ma YS, Xiao LK. Postoperative Pain Management in Total Knee Arthroplasty. Orthop Surg. 2019 Oct;11(5):755-761. doi: 10.1111/os.12535. PMID 31663286
- [Background] Horlocker TT. Pain management in total joint arthroplasty: a historical review. Orthopedics. 2010 Sep;33(9 Suppl):14-9. doi: 10.3928/01477447-20100722-65. PMID 20839717
- [Background] Soffin EM, Memtsoudis SG. Anesthesia and analgesia for total knee arthroplasty. Minerva Anestesiol. 2018 Dec;84(12):1406-1412. doi: 10.23736/S0375-9393.18.12383-2. Epub 2018 May 28. PMID 29808972
- [Background] Pugely AJ, Martin CT, Gao Y, Mendoza-Lattes S, Callaghan JJ. Differences in short-term complications between spinal and general anesthesia for primary total knee arthroplasty. J Bone Joint Surg Am. 2013 Feb 6;95(3):193-9. doi: 10.2106/JBJS.K.01682. PMID 23269359